CLINICAL TRIAL: NCT01086293
Title: Comparison of Risk of Hospitalization With Acute Liver Failure Between Patients With Type 2 Diabetes Initiating Saxagliptin and Those Initiating Other Oral Antidiabetic Treatments
Brief Title: Risk of Acute Liver Failure Among Patients With Type 2 Diabetes Exposed to Oral Antidiabetic Treatments
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: CV181-100
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients exposed to Saxagliptin
- Patients exposed to oral antidiabetic drugs (not Saxagliptin)

SUMMARY:
The purpose of this study is to compare the incidence of hospitalization with acute liver failure among patients with type 2 diabetes who are new users of Saxagliptin and those who are new users of other oral antidiabetic drugs.

DETAILED DESCRIPTION:
Prospectively designed retrospective database study. This study will be conducted using administrative claims data and electronic medical records that are collected as part of routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Newly prescribed Saxagliptin or an Oral Antidiabetic Drug (OAD) in a class other than Dipeptidyl peptidase IV (DPP4) inhibitors
* Enrolled in the respective database for at least 180 days prior to the first prescription of new OAD
* Have at least one diagnostic code for a type 2 diabetes-related condition

Exclusion Criteria:

* Patients identified with a diagnostic code for acute liver failure within the 180-day baseline period
* Patients with DPP4 inhibitor exposure during the baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out using databases containing administrative claims data (HealthCore Integrated Research DatabaseSM (HIRD) and Medicare in the U.S.) and electronic medical records (General Practice Research Database (GPRD) and The Health Improvement Network (THIN) in the UK). The US population includes patients from health plans in the northeast, southeastern, mid-Atlantic, central, mid-western, and western regions (HIRD) as well as US citizens 65 years of age and older (Medicare). The UK population includes patients seeking medical care from general practitioners (GPRD and THIN)
Sampling Method: Non-Probability Sample
Enrollment: 113505 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants hospitalized with a diagnosis of acute liver failure | 18-months
Number of participants hospitalized with a diagnosis of acute liver failure | 36-months
Number of participants hospitalized with a diagnosis of acute liver failure | 54-months

SECONDARY OUTCOMES:
Deaths due to acute liver failure | 18, 36 and 54 months
Hospitalizations with acute liver failure and/or death due to acute liver failure | 18, 36 and 54 months
Hospitalizations with acute liver injury | 18, 36 and 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Lo Re V, Carbonari DM, Saine ME, Newcomb CW, Roy JA, Liu Q, Wu Q, Cardillo S, Haynes K, Kimmel SE, Reese PP, Margolis DJ, Apter AJ, Reddy KR, Hennessy S, Bhullar H, Gallagher AM, Esposito DB, Strom BL. Postauthorization safety study of the DPP-4 inhibitor saxagliptin: a large-scale multinational family of cohort studies of five outcomes. BMJ Open Diabetes Res Care. 2017 Jul 31;5(1):e000400. doi: 10.1136/bmjdrc-2017-000400. eCollection 2017. PMID 28878934
- [Derived] Saine ME, Carbonari DM, Newcomb CW, Nezamzadeh MS, Haynes K, Roy JA, Cardillo S, Hennessy S, Holick CN, Esposito DB, Gallagher AM, Bhullar H, Strom BL, Lo Re V 3rd. Determinants of saxagliptin use among patients with type 2 diabetes mellitus treated with oral anti-diabetic drugs. BMC Pharmacol Toxicol. 2015 Apr 2;16:8. doi: 10.1186/s40360-015-0007-z. PMID 25889498
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4451&filename=cv181_100.pdf